CLINICAL TRIAL: NCT02317289
Title: Development of a Multimodal Controlled Device for Improvement and Monitoring of Freezing in Parkinsonian Patients
Brief Title: Assisted Device for Freezing in Parkinson Disease
Acronym: demarpark
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period and recruitment difficulties
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9096
Record Dates: First submitted 2014-12-03; First posted 2014-12-15 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Detection of freezing (Experimental): freezing parkinsonian patients
  Interventions: Device: Detection of freezing

INTERVENTIONS:
Device: Detection of freezing — single wireless inertial sensor placed on the patients's lower limbs to detect freezing of gaitin Parkinsonian patients
  Other Names: SENSBIO

SUMMARY:
Freezing of gait (FOG) is a particular and troublesome symptom occurring in some Parkinsonian patients. Our objective is to adapt and extend FOG detectors in order to include other associated gait pattern changes, like festination.Our purpose is to develop a wearable assistant which would trigger the most appropriate cueing aid just before occurrence of the freezing episode.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is a particular and troublesome symptom occurring in some Parkinsonian patients .This brief, episodic absence or marked reduction of forward progression of the feet despite the intention to walk is associated to a fall risk. Automatized FOG episode detection would allow systematic assessment of patient state and objective evaluation of the clinical effects of treatments. Techniques have been proposed in the literature to identify FOG episodes based on the frequency properties of inertial sensor signals. Our objective here is to adapt and extend these FOG detectors in order to include other associated gait pattern changes, like festination. The proposed approach is based on a single wireless inertial sensor placed on the patient's lower limbs. Based freezing detectors are not sufficient to detect all FOG and festination episodes. Stride length and cadence are valuable inputs to anticipate the occurrence of upcoming FOG events. The investigators have developed a solution based on a minimal number of embedded sensors and detection algorithms for future real-time applications. It is well known that auditory rhythmic stimulation or visuals marks on the ground would improve dramatically gait in patients with FOG. This sensibility to cueing leads some teams to develop some mobility aid devices rhythmic. Our purpose is to develop a wearable assistant which would trigger the most appropriate cueing aid just before occurrence of the freezing episode.

ELIGIBILITY:
Inclusion Criteria:

* troublesome freezing

Exclusion Criteria:

* dementia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2015-10-13 (Actual)

PRIMARY OUTCOMES:
fog score | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Christian GENY, MD, Principal Investigator — CHRU Montpellier
Locations (1):
- Gui de Chauliac Hospital, Montpellier, France